CLINICAL TRIAL: NCT01575275
Title: A Phase 2 Comparative Study of 5-Aminolevulinic Acid (5-ALA) and Intraoperative MRI (iMRI) to Enhance Completeness of Resection of Glioblastoma
Brief Title: Aminolevulinic Acid in Visualizing a Tumor During Surgery in Patients With Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: Michael Vogelbaum, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Vogelbaum, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE1311; NCI-2012-00452 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (aminolevulinic acid) (Experimental): Patients receive aminolevulinic acid PO 2-4 hours before surgery.
  Interventions: Drug: aminolevulinic acid; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: aminolevulinic acid — Given PO
  Other Names: 5-ALA; 5-Aminolaevulinic Acid; ALA
Procedure: therapeutic conventional surgery — Undergo surgery

SUMMARY:
The purpose of this study is to investigate the safety and performance of an investigational agent, known as 5-ALA or Gliolan (aminolevulinic acid), that many be useful to a surgeon for visualizing a tumor during surgery. It is also being studied to determine if there are differences in what Gliolan shows a surgeon compared to intraoperative magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the volume of residual enhancing tumor after a 5-ALA guided resection of a glioblastoma multiforme (GBM).

II. Determine the volume of tissue removed compared to the measured enhancing tumor evaluated on a pre-operative MRI.

SECONDARY OBJECTIVES:

I. Evaluate the time to tumor progression. II. Evaluate the overall survival.

OUTLINE:

Patients receive aminolevulinic acid orally (PO) 2-4 hours before surgery.

After completion of study treatment, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a suspected or biopsy proven newly diagnosed GBM, or a recurrent GBM or suspected GBM (in patient with pathologically diagnosed prior World Health Organization [WHO] grade II or III tumor) in a patient undergoing a clinically-indicated surgery.
* Age >= 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy is not a consideration for protocol entry
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits; OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document or have a parent or guardian with the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Prior therapy is not an exclusion criterion
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to aminolevulinic acid (ALA)
* Current treatment with hypericin (or an extract) or other photosensitizing agents
* Personal or immediate family (parents, siblings, children) history of porphyrias
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ALA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vogelbaum, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Aminolevulinic Acid)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Aminolevulinic Acid)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Volume of Residual Enhancing Tumor, as Determined by Intraoperative Volume MRI at a Single Time Point Without and With Gadolinium, Following Maximal Resection With Use of Aminolevulinic Acid
Description: Volume of enhancing tumor (initial and residual) will be determined by use of a softwarebased volumetric analysis method. Intra- and post-op definitions of residual tumor volume need to be adjusted for the presence of T1 hyperintensity due to signal from blood and blood products (as determined on pre-gadolinium volume study).
Time Frame: Day 1
Measure: Median (Full Range); unit: cc
Arm/Group | Diagnostic (Aminolevulinic Acid)
Number analyzed (Participants) | 8
cc | -0.342 [-2.604 to 1.096]

2. Primary Outcome: Comparison Between the Volume of Resected Tissue (Defined as the Volume of the Resection Cavity) and the Pre-operative Enhancing Tumor Volume
Description: Volume of enhancing tumor (initial and residual) will be determined by use of a software-based volumetric analysis method. Intra- and post-op definitions of residual tumor volume need to be adjusted for the presence of T1 hyperintensity due to signal from blood and blood products (as determined on pre-gadolinium volume study).
Time Frame: Up to day 1
Population: Outcome never analyzed. Study closed with the IRB in 2014
Arm/Group | Diagnostic (Aminolevulinic Acid)
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Disease Progression (TTP), Determined by Review of MRIs Performed Post Operatively as Clinically Indicated, Evaluated With Use of the New International Criteria Proposed by the Response in NeuroOncology (RANO) Committee
Time Frame: From the date of surgery with aminolevulinic acid to the date of progression, assessed up to 1 year
Population: Outcome never analyzed. Closed with the IRB in 2014
Arm/Group | Diagnostic (Aminolevulinic Acid)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival, by Periodic Follow up Review of the Patient Charts and by Correlation With the Social Security Death Index
Time Frame: From the date of surgery with aminolevulinic acid to the date of death, assessed up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Diagnostic (Aminolevulinic Acid)
Number analyzed (Participants) | 8
months | 16 [8 to 38]

ADVERSE EVENTS:
Arm/Group | Diagnostic (Aminolevulinic Acid)
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Aminolevulinic Acid) (N=8)
Infection (Nervous system disorders) | 1 (1) — Meningitis
Syncope (Cardiac disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Aminolevulinic Acid) (N=8)
hypoalbuminemia (Investigations) | 2 (3)
Hypocalcemia (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Infection with unknown ANC - Meninges (Infections and infestations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neuropathy: Sensory (Nervous system disorders) | 1 (1)
Pain (General disorders) | 2 (6)
Low Platelets (Blood and lymphatic system disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
hyponatremia (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No